CLINICAL TRIAL: NCT02990715
Title: Evaluation of Check-Cap C-Scan System in Providing Structural Information and Detection of Polypoid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CL-SY-01-0093
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Polypoid Lesions
Keywords: average risk CRC screening; Non compliant patients for CRC screening; Counterindicated patients for colonoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The colonoscopists will be blinded to the C-Scan system results and FIT results and the reviewers of C-Scan system results will be blinded to Fit and colonoscopy results

ARMS (2):
- Up to 45 subjects (Active Comparator): Subjects with known polyp lesions≥10mm which were not removed because of poor preperation or the need to perform polypectomy at hospital will ingest the C-Scan cap and then will be schduled to polypectomy. The subjects will perform FIT test during the procedure and it will be compared with C-Scan System results.
  Interventions: Device: C-Scan System
- Up to 25 subjects (Experimental): Subjects who were reffered to screening colonoscopy as an average risk for CRC will ingest the C-Scan cap and then will be schduled to polypectomy. The subjects will perform FIT test during the procedure and it will be compared with C-Scan System results.
  Interventions: Device: C-Scan System

INTERVENTIONS:
Device: C-Scan System — 1. To establish the efficacy of C-Scan Capsule System and FIT in detecting patients with polypoid lesions ≥ 10mm, compared with Optical Colonoscopy
  2. To evaluate the safety of the C-Scan Capsule System procedure
  Other Names: Colon capsule

SUMMARY:
The purpose of this study is to establish the efficacy of Check-Cap's C-Scan System in providing structural information on colonic polypoid lesions and masses, as an adjacent tool to FIT.

DETAILED DESCRIPTION:
The subject will be invited to come to the clinic to sign the ICF and other related documents. Then they'll ingest the capsule typically during the morning hours. The subjects will be connected to the C-Scan Track and system's activation the subject will be asked to ingest the C-Scan Capsule with some water and contrast media, in the presence of a physician.

Post ingestion, the subject will be discharged home with clear instructions on the procedure. The subject should avoid intensive physical exercise during procedure or any extreme activities. The subject should make an effort to stay at home or other familiar surroundings, and may continue daily activities such mobile/computer/TV use, shower, sleep or eat. Details on allowed and restricted activities are listed in app. 4 The subject will be required to ingest daily dose (3 X 15-17ml) of contrast media, to be consumed three times per day with normal diet. Also on a need based the subject would be provided with laxadine (5 mg tablets) to be ingested according to the doctor recommendation.

During capsule procedure the subjects will be contacted by phone several times daily by the site clinical study team (or by dedicated external trained medical personnel), to assure the subjects well-being and to monitor for any change or discomfort and for procedure progress. Subjects may be also monitored by the technical team (either at home or at the clinic), who may need to examine the system or inquire the subjects about the system visual/auditory indicators.

The subjects will be provided with a dedicated capsule collection kit, to assist the subjects in collecting the capsule. Subjects will be instructed to retrieve the capsule upon excretion.

Capsule procedure is completed upon capsule excretion or system vibro/auditory indication of 'End of Procedure'.

Patients will be instructed to return the C-Scan Capsule and C-Scan Track to the clinic for analysis.

All subjects will be scheduled for optical colonoscopy to be performed within one month following capsule procedure.

C-Scan Procedure Analysis:

Two to three licensed gastroenterologist physicians, will be trained with reviewing and analyzing C-Scan System scans, to serve as independent reviewers. A reviewing forum consisting of at least one independent trained gastroenterologist physician and at least 2 expert Check-Cap reviewers that will jointly review all the cases. The reviewing forum will be blinded to the FIT and colonoscopy results of the examined patients..). Analysis will be performed on a per patient basis for the existence or non-existence of a finding that may be a polyp. This per patient finding will be compared with the FIT, and a colonoscopy will be performed for verification.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at the age of 30-80 years old
* Subject provided signed informed consent

Exclusion Criteria:

* Patients with advanced cancer or other life threatening diseases or conditions
* Subject with known history of dysphagia or other swallowing disorders
* Subject with known history of GI disease or symptoms, such as: Crohn's disease, Colitis, IBD, Meckel's Diverticulum, Bowen Hernia, Mega Colon, fistulas or other strictures (doctors' discretion).
* Subject with known motility disorder or Chronic Constipation
* Subject with known delayed gastric emptying
* Subject with prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by physician discretion
* Subject with any condition believed to have an increased risk for capsule retention such as intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy, as determined by physician discretion
* Subject with a cardiac pacemaker or other implanted electro medical device
* Subjects with known sensitivity to iodine, or with kidney failure
* Subjects with morbid obesity (BMI > 40)
* Subject with any known condition which precludes compliance with study and/or device instructions
* Subject with known condition of drug abuse and/or alcoholism
* Subject who is unable to undergo colonoscopy or bowel preparation necessary for colonoscopy (based on previous attempts or self-declaration)
* Women who are either pregnant or nursing at the time of screening (to be verified by test in case of woman of child-bearing potential that do not practice medically acceptable methods of contraception)
* Concurrent participation in another clinical trial using any investigational drug or device

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09-10 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of C-Scan Capsule System in detecting per segment polypoid lesions 10 mm and up as compared with Colonoscopy | One year
  Number of polyps detected by the capsulle system in variuos segements of the colon as compared with the results indicated in the report of the follow-up colonoscopy

SECONDARY OUTCOMES:
Sensitivity and specificity of C-Scan Capsule System in detecting patients with polypoid lesions 6≤x≤9 mm, compared with Optical Colonoscopy | One year
  Number of polyp specificity of C-Scan Capsule System in detecting patients with polypoid lesions 6≤x≤9 mm detected by the capsule system in variuos segements of the colon as

CONTACTS AND LOCATIONS:
Overall Officials: Alex Ovadia, Study Director — COO, VP R&D
Locations (3):
- Israel (3):
  - Emek Medical Center, Afula, Galilee
  - Rambam Medical Center, Haifa, North
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
Preliminary results will be presented in the European Gatro Conference UEGW on October 2017